CLINICAL TRIAL: NCT05064761
Title: A Pilot Study to Evaluate Safety and Effectiveness of Poly-l-lactic Acid (PLLA) for the Improvement in Appearance of Cellulite
Brief Title: Safety and Effectiveness of Poly-l-lactic Acid (PLLA) for the Improvement in Appearance of Cellulite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 43CASA2006
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Results first posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-05

CONDITIONS: Cellulite
MeSH Terms: conditions — Cellulite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment group (Experimental): PLLA new dilution for treatment to improve appearance of cellulite.
  Interventions: Device: Sculptra new dilution

INTERVENTIONS:
Device: Sculptra new dilution — Treatment to improve appearance of cellulite.

SUMMARY:
This pilot study has been designed to evaluate the safety and effectiveness of PLLA as a single regimen for the improvement in appearance of cellulite after changes in reconstitution procedure.

DETAILED DESCRIPTION:
Cellulite is a topographic and localized skin condition that is commonly found on the posterolateral thighs, buttocks, and abdomen. It is often identified by a dimpled or orange-peel appearance of the skin's surface. The presence of visible cellulite is associated with histologic changes in the dermis, adipose tissue, and septae.

Based on the theory that a stronger skin structure, with a decrease in skin laxity and increase in dermal thickness, could reduce the appearance of cellulite, the Sponsor intends to investigate the safety and effectiveness of PLLA for the improvement in appearance of cellulite in the posterior thighs.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with intent to undergo treatment to improve appearance of cellulite in the posterior thighs.

Exclusion Criteria:

* Known/previous allergy or hypersensitivity to any of the Sculptra constituents.
* Known/previous allergy or hypersensitivity to lidocaine and other local anesthetics, e.g. amide-type anesthetics, or topical anesthetics or nerve blocking agents.
* Previous or present multiple allergies or severe allergies, such as manifested by anaphylaxis or angioedema, or family history of these conditions.
* Previous treatment/procedure in or near the treatment area:

  1. Previous permanent implant, filler, lifting threads, or autologous fat in the treatment area, regardless of time.
  2. Previous semi-permanent implants exemplified by Calcium Hydroxylapatite (CaHA), poly l-lactic acid (PLLA) in treatment area, regardless of time.
  3. Previous Hyaluronic acid (HA) filler or collagen filler in the treatment area within 12 months.
  4. Previous energy based aesthetic procedures (e.g. laser, intense pulsed light, radiofrequency and endermology) in the treatment area within 6 months.
  5. Previous mechanical (e.g. dermabrasion, needling) or chemical aesthetic procedures (e.g. chemical peel) in the treatment area within 6 months.
  6. Previous treatment with cryotherapy, lipolytic treatments or liporeduction massage in the treatment area within 6 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2023-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Galderma R&D
Locations (1):
- Galderma Research Site, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at Canada from 19 November 2021 to 27 February 2023.
Pre-assignment Details: A total of 29 participants were enrolled in the study. All enrolled participants were treated and completed the study.
Groups:
- Treatment Group (Sculptra): Participants with intent to undergo treatment to improve appearance of cellulite were enrolled and treated with Sculptra in three sessions spaced one month (+2 weeks) apart. Participants were treated at baseline, Month 1 and Month 2.
Period: Overall Study
Arm/Group | Treatment Group (Sculptra)
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Group (Sculptra)
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (9.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Aesthetic Improved Thighs of Responders According to Global Aesthetic Improvement Scale (GAIS) as Assessed Live by Treating Investigator at Month 9
Description: Aesthetic improvement was assessed by comparing a photograph taken before the first treatment at the baseline visit to current visit. On a 7-graded GAIS from "very much worse" to "very much improved" as follows; very much improved, much improved, improved, no change, worse, much worse and very much worse. Responder was defined as a participant with a rating of at least improved as assessed by the treating investigator (assessed as very much improved, much improved or improved) compared to pre-treatment. Number of aesthetic improved thighs of responders based on treating investigator assessment using GAIS at Month 9 were reported.
Time Frame: At Month 9
Population: Full Analysis Set (FAS) Included all participants who were injected in both thighs.
Measure: Count of Units; unit: Thighs
Units Other Than Participants: Thighs
Arm/Group | Treatment Group (Sculptra)
Number analyzed (Participants) | 29
Number analyzed (Thighs) | 58
Thighs
  Left thigh: number analyzed (Thighs) | 29
  Left thigh: Very much improved | 23
  Left thigh: Much improved | 4
  Left thigh: Improved | 1
  Left thigh: No change | 1
  Right thigh: number analyzed (Thighs) | 29
  Right thigh: Very much improved | 24
  Right thigh: Much improved | 3
  Right thigh: Improved | 1
  Right thigh: No change | 1

2. Secondary Outcome: Number of Aesthetic Improved Thighs of Responders According to Global Aesthetic Improvement Scale (GAIS) as Assessed Live by Treating Investigator at Month 1, 2, 6 and 12
Description: Aesthetic improvement was assessed by comparing a photograph taken before the first treatment at the baseline visit to a photograph from the current visit. on a 7-graded GAIS from "very much worse" to "very much improved" as follows; very much improved, much improved, improved, no change, worse, much worse and very much worse. Responder was defined as a participant with a rating of at least improved as assessed by the treating investigator (assessed as very much improved, much improved or improved) compared to pre-treatment. Number of aesthetic improved thighs of responders based on treating investigator assessment using GAIS at Month 1,2,6 and 12 were reported.
Time Frame: At month 1, 2, 6 and 12
Population: Full Analysis Set (FAS) Included all participants who were injected in both thighs.
Measure: Count of Units; unit: Thighs
Units Other Than Participants: Thighs
Arm/Group | Treatment Group (Sculptra)
Number analyzed (Participants) | 29
Number analyzed (Thighs) | 58
Thighs
  Month 1, Left thigh: number analyzed (Thighs) | 29
  Month 1, Left thigh: Very much improved | 0
  Month 1, Left thigh: Much improved | 8
  Month 1, Left thigh: Improved | 16
  Month 1, Left thigh: No change | 5
  Month 1, Right thigh: number analyzed (Thighs) | 29
  Month 1, Right thigh: Very much improved | 1
  Month 1, Right thigh: Much improved | 6
  Month 1, Right thigh: Improved | 17
  Month 1, Right thigh: No change | 5
  Month 2, Left thigh: number analyzed (Thighs) | 29
  Month 2, Left thigh: Very much improved | 2
  Month 2, Left thigh: Much improved | 8
  Month 2, Left thigh: Improved | 19
  Month 2, Left thigh: No change | 0
  Month 2, Right thigh: number analyzed (Thighs) | 29
  Month 2, Right thigh: Very much improved | 2
  Month 2, Right thigh: Much improved | 8
  Month 2, Right thigh: Improved | 19
  Month 2, Right thigh: No change | 0
  Month 6, Left thigh: number analyzed (Thighs) | 29
  Month 6, Left thigh: Very much improved | 16
  Month 6, Left thigh: Much improved | 7
  Month 6, Left thigh: Improved | 6
  Month 6, Left thigh: No change | 0
  Month 6, Right thigh: number analyzed (Thighs) | 29
  Month 6, Right thigh: Very much improved | 16
  Month 6, Right thigh: Much improved | 6
  Month 6, Right thigh: Improved | 7
  Month 6, Right thigh: No change | 0
  Month 12, Left thigh: number analyzed (Thighs) | 29
  Month 12, Left thigh: Very much improved | 18
  Month 12, Left thigh: Much improved | 10
  Month 12, Left thigh: Improved | 1
  Month 12, Left thigh: No change | 0
  Month 12, Right thigh: number analyzed (Thighs) | 29
  Month 12, Right thigh: Very much improved | 19
  Month 12, Right thigh: Much improved | 8
  Month 12, Right thigh: Improved | 2
  Month 12, Right thigh: No change | 0

3. Secondary Outcome: Number of Aesthetic Improved Thighs of Responders According to Global Aesthetic Improvement Scale (GAIS) as Assessed by Participant Photography at Month 1, 2, 6, 9 and 12
Description: Aesthetic improvement was assessed by comparing a photograph taken before the first treatment at the baseline visit to a photograph from the current visit. on a 7-graded GAIS from "very much worse" to "very much improved" as follows; very much improved, much improved, improved, no change, worse, much worse and very much worse. Responder was defined as a participant with a rating of at least improved as assessed by themselves (assessed as very much improved, much improved or improved) compared to pre-treatment. Number of aesthetic improved thighs of responders based on participant photography assessment using GAIS at Month 1,2,6 and 12 were reported.
Time Frame: At Months 1, 2, 6, 9 and 12
Population: Full Analysis Set (FAS) Included all participants who were injected in both thighs. Here, "Number analyzed" signifies those units (thighs) which were evaluable at the specified timeframe.
Measure: Count of Units; unit: Thighs
Units Other Than Participants: Thighs
Arm/Group | Treatment Group (Sculptra)
Number analyzed (Participants) | 29
Number analyzed (Thighs) | 58
Thighs
  Month 1, Left thigh: number analyzed (Thighs) | 29
  Month 1, Left thigh: Very much improved | 2
  Month 1, Left thigh: Much improved | 3
  Month 1, Left thigh: Improved | 19
  Month 1, Left thigh: No change | 5
  Month 1, Right thigh: number analyzed (Thighs) | 29
  Month 1, Right thigh: Very much improved | 2
  Month 1, Right thigh: Much improved | 2
  Month 1, Right thigh: Improved | 20
  Month 1, Right thigh: No change | 5
  Month 2, Left thigh: number analyzed (Thighs) | 29
  Month 2, Left thigh: Very much improved | 5
  Month 2, Left thigh: Much improved | 8
  Month 2, Left thigh: Improved | 14
  Month 2, Left thigh: No change | 2
  Month 2, Right thigh: number analyzed (Thighs) | 29
  Month 2, Right thigh: Very much improved | 4
  Month 2, Right thigh: Much improved | 9
  Month 2, Right thigh: Improved | 14
  Month 2, Right thigh: No change | 2
  Month 6, Left thigh: number analyzed (Participants) | 28
  Month 6, Left thigh: number analyzed (Thighs) | 28
  Month 6, Left thigh: Very much improved | 6
  Month 6, Left thigh: Much improved | 9
  Month 6, Left thigh: Improved | 11
  Month 6, Left thigh: No change | 2
  Month 6, Right thigh: number analyzed (Participants) | 28
  Month 6, Right thigh: number analyzed (Thighs) | 28
  Month 6, Right thigh: Very much improved | 6
  Month 6, Right thigh: Much improved | 8
  Month 6, Right thigh: Improved | 13
  Month 6, Right thigh: No change | 1
  Month 9, Left thigh: number analyzed (Thighs) | 29
  Month 9, Left thigh: Very much improved | 11
  Month 9, Left thigh: Much improved | 5
  Month 9, Left thigh: Improved | 11
  Month 9, Left thigh: No change | 2
  Month 9, Right thigh: number analyzed (Thighs) | 29
  Month 9, Right thigh: Very much improved | 11
  Month 9, Right thigh: Much improved | 5
  Month 9, Right thigh: Improved | 12
  Month 9, Right thigh: No change | 1
  Month 12, Left thigh: number analyzed (Thighs) | 29
  Month 12, Left thigh: Very much improved | 12
  Month 12, Left thigh: Much improved | 5
  Month 12, Left thigh: Improved | 10
  Month 12, Left thigh: No change | 2
  Month 12, Right thigh: number analyzed (Thighs) | 29
  Month 12, Right thigh: Very much improved | 11
  Month 12, Right thigh: Much improved | 6
  Month 12, Right thigh: Improved | 10
  Month 12, Right thigh: No change | 2

ADVERSE EVENTS:
Time Frame: Up to 12 months
Arm/Group | Treatment Group (Sculptra)
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 10/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group (Sculptra) (N=29)
Bronchitis (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Urethral prolapse (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-21): https://cdn.clinicaltrials.gov/large-docs/61/NCT05064761/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-29): https://cdn.clinicaltrials.gov/large-docs/61/NCT05064761/SAP_001.pdf